CLINICAL TRIAL: NCT06320678
Title: Effect of Concept Mapped Blended Learning Self-Directed Learning on the Knowledge Level of Parenteral Drug Administration in Nursing Students: a Randomized Controlled Study
Brief Title: Parenteral Drug Administration Training for Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Aysun Acun 5
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-02

CONDITIONS: Nursing Education
Keywords: Concept Map; Blended Learning; Nursing Students; Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blended Learning (Experimental)
  Interventions: Other: Nursing Students Education
- Education (No Intervention)

INTERVENTIONS:
Other: Nursing Students Education — Effect of Concept Mapped Blended Learning Self-Directed Learning
  Arms: Blended Learning

SUMMARY:
This study aims to evaluate the effect of blended self-directed learning with concept mapping on the level of knowledge regarding parenteral drug administration in nursing students. With out-of-class, online, interactive teaching methods, a memorable learning away from complex structure is aimed.

DETAILED DESCRIPTION:
Online learning materials are of great importance in health education where theoretical knowledge and psychomotor skills are developed. The student takes responsibility for learning and has the chance to continue his education outside the classroom. Concept maps are one of the most effective educational materials both in classroom education and online learning. Visual education is concept map training in which each concept is included once on concrete applications and the relationships between concepts are revealed within the framework of the main lines to be taught. Providing parenteral drug administration training with a concept map will reveal the application steps as a concrete step and clear away confusing theoretical knowledge. The use of concept maps will ensure that first-year nursing students who are receiving training on drug administration for the first time will receive an education that is summative and memorable, away from the complex structure. One of the education models that offer interactive education opportunities other than traditional ones is blended learning. Blended learning provides a combination of face-to-face and technology-mediated teaching and learning that not only fully embodies the concept of "student-centered" teaching but also enables students to effectively participate in the classroom. The student-centered nature of blended learning also brings about self-directed learning. Self-directed learning is defined as the process of constantly monitoring and improving students' cognitive states, observing and applying various learning strategies, helping them recognize learning behaviors, and making efforts to create and use physical and social resources that facilitate learning.

ELIGIBILITY:
Inclusion Criteria:

* Receiving Parenteral Drug Administration training for the first time
* Becoming a first-year nursing student
* Volunteering to participate in research

Exclusion Criteria:

* Not participating in posttest and follow-up tests
* Not volunteering to participate in the research

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Students' knowledge level after blended learning method | 5 week
  Students' learning of parenteral drug administration will be examined with the blended learning method.

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Bilecik, Turkey (Türkiye)